CLINICAL TRIAL: NCT01315613
Title: Study of ST2-IL-33 Pathway in Acute Pancreatitis
Brief Title: Role of ST2 in Acute Pancreatitis
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Romy Ouziel,, Erasme Hospital
Other Study IDs: RO-ST2
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2008-09

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Acute pancreatitis: Patients admitted in our institution for an episode of acute pancreatitis

SUMMARY:
Acute pancreatitis is characterized by an inflammatory storm which regulatory pathways are not well known. The IL-1 cytokine family is activated early during acute pancreatitis and secretion of alarmins is speculated during pancreatic necrosis. IL-33 is a member of the IL-1 family, it can act as an alarmin and its receptor, ST2, is known to sequester MyD88 which might regulate the acute pancreatitis inflammatory storm. The aim of this study is to investigate ST2 pathway in human acute pancreatitis and in murine experimental models of acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Time to take blood sample less than 24h after the onset of symptoms of AP
* Two of the following: typical pain, amylase and lipase concentrations more than 3x the upper normal limit, compatible modifications on imaging techniques

Exclusion Criteria:

* Chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of Erasme University Hospital
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09

PRIMARY OUTCOMES:
Concentration of soluble ST2 in serum | Within 30 days after onset of acute pancreatitis
  Concentration of soluble ST2 will be assessed in the serum of patient with an episode of acute pancreatitis, on the day of admission to the hospital as well as 24h, 48h, 7 days and 30 days later.

CONTACTS AND LOCATIONS:
Overall Officials: Romy Ouziel, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme Hospital, Brussels, Belgium